CLINICAL TRIAL: NCT07064369
Title: Observational Study on the Clinical, Laboratory, Anatomopathological, and Molecular Characteristics and Their Prognostic and Predictive Value in Patients With Thyroid Tumors Treated at the Fondazione Policlinico Universitario A.Gemelli IRCCS.
Brief Title: Observational Study on Thyroid Tumors and EvaLuation of the roLe of New pOntential Predictive/Prognostic Factors
Acronym: OTELLO
Status: Enrolling by invitation | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6506
Record Dates: First submitted 2025-02-07; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-02

CONDITIONS: Carcinoma of Head/Neck
Keywords: thyroid; thyroid carcinoma
MeSH Terms: conditions — Thyroid Diseases; Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Historical (Retrospective) Cohort: The medical records of patients diagnosed with thyroid neoplasms and followed at the Medical Oncology Unit of the Fondazione Policlinico Universitario Agostino Gemelli (FPG) - IRCCS from January 1, 2010, until the date of study approval will be screened for retrospective analysis.
  Cases that meet the inclusion and exclusion criteria will be selected, and their medical records will be reviewed by the investigators to collect the required information.
  For patients who are still alive, they will be contacted to discuss the study and, if they agree to participate, they will be asked to sign the informed consent (IC) and the data privacy consent form
- Prospective Cohort: Patients diagnosed with thyroid neoplasms who present to the Medical Oncology Unit of the Fondazione Policlinico Universitario Agostino Gemelli (FPG) - IRCCS after the protocol approval date and within the following 60 months will be screened.
  If they meet the inclusion and exclusion criteria, they will be enrolled in the study after signing the informed consent (IC) and the data privacy consent form.

SUMMARY:
The OTELLO Study is a monocentric, ambispective observational study that systematically analyzes the clinical, laboratory, anatomopathological, and molecular characteristics of patients with thyroid neoplasms treated at the Agostino Gemelli University Hospital - IRCCS.

Study Objectives

The primary goal is to identify prognostic and predictive factors that can enhance the clinical and therapeutic management of thyroid cancer patients at any disease stage. The analysis aims to integrate biological tumor characteristics with clinical and therapeutic data to identify significant correlations between these parameters and disease progression.

Study Design and Patient Cohorts

The study includes two distinct cohorts:

Historical (retrospective) cohort: This group includes patients previously treated for thyroid neoplasms from January 1, 2010, to the date of study approval. Data from these patients will be analyzed to evaluate long-term outcomes and identify potential predictors of treatment response.

Prospective cohort: This group includes patients newly diagnosed with thyroid cancer who will be enrolled over a 60-month period from the study's approval. These patients will undergo systematic monitoring to assess disease progression and therapy effectiveness.

Data Collection and Analysis

The study will collect and examine data on:

Clinical characteristics: Including sex, age at diagnosis, comorbidities, hereditary syndromes, and performance status.

Laboratory data: Including tumor markers and metabolic parameters relevant to disease characterization.

Anatomopathological aspects: Such as histological tumor type, pathological staging, lymphovascular or perineural invasion, and other indicators of tumor aggressiveness.

Molecular profiles: Evaluated through genetic alterations and biomarkers with potential prognostic and predictive value.

Statistical and Methodological Approach

An advanced statistical approach will be used to assess the impact of collected variables on patient outcomes. The analysis will include:

Comparative analyses of patient groups based on clinical and biological characteristics.

Survival analysis, estimating overall survival (OS) and progression-free survival (PFS) using Kaplan-Meier curves and log-rank tests.

Multivariate regression models to identify independent factors associated with prognosis and treatment response.

Ethical Considerations and Regulatory Compliance

The study will be conducted in compliance with ethical and regulatory guidelines, including the Declaration of Helsinki, Good Clinical Practice (GCP) by ICH, and Italian regulations on observational studies. Patient data will be anonymized and securely stored, ensuring confidentiality.

As a non-interventional study, no experimental drugs or procedures will be administered. However, molecular and immunohistochemical analyses will be performed on tumor tissue samples already available or collected during standard clinical practice.

Study Timeline and Expected Outcomes

The prospective cohort enrollment will continue until 2029, after which statistical analyses will be completed, and study results will be published. The collected data will provide valuable insights for optimizing the clinical management of thyroid cancer patients, supporting the development of increasingly personalized diagnostic and therapeutic strategies.

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE OF THE STUDY

Thyroid tumors are the most common endocrine malignancies worldwide. Due to improved diagnostic techniques and increased adherence to screening procedures, incidence rates are rising [1]. In Italy, thyroid cancer is approximately three times more frequent in women (23.6 per 100,000 per year in 2003-2014) than in men (8.4 per 100,000 per year) [2]. Among the main histological types, approximately 90% are papillary thyroid carcinomas (PTC), 4% are follicular thyroid carcinomas (FTC), 2% are Hürthle cell carcinomas, 2% are medullary thyroid carcinomas (MTC), and 1% are anaplastic thyroid carcinomas (ATC) [3].

MTCs are neuroendocrine tumors arising from calcitonin-producing C cells (parafollicular cells). Other rare thyroid tumors, with some exceptions (e.g., squamous carcinoma, lymphoma, mesenchymal tumors), originate from follicular cells. Well-differentiated thyroid cancer (DTC) accounts for about 95% of thyroid malignancies, with 5% of these cases being familial. Most familial thyroid cancer cases are non-medullary (NMFTC) and occur within complex familial syndromes such as familial adenomatous polyposis (FAP), Cowden syndrome, Carney complex, Pendred syndrome, and Werner syndrome [4]. Familial cases of PTC, FTC, and ATC are rare, accounting for only 5% of cases (mainly in PTC patients). Conversely, MTC is inherited as an autosomal dominant trait in 25% of cases, whereas 75% of MTC cases are sporadic, with somatic mutations in RET, followed by H-RAS and K-RAS [5].

Hereditary MTC associated with RET mutations falls under the multiple endocrine neoplasia type 2 (MEN2) syndrome, further classified into three subtypes based on clinical phenotype (MEN2A, MEN2B, and familial medullary thyroid carcinoma (FMTC)) [6]. Beyond germline mutations, the 2014 Cancer Genome Research Network identified driver somatic mutations in over 95% of PTCs [7,8], including BRAF mutations (especially BRAFV600), TERT promoter mutations (often coexisting), and RAS mutations. These mutations are also implicated in the early molecular events leading to poorly differentiated and anaplastic thyroid carcinomas, alongside TP53 mutations, which contribute to PTC progression [5].

The detection of these genomic alterations has significant prognostic [5,9] and therapeutic implications. Additionally, RET/PTC rearrangements are another hallmark molecular event, frequently observed in PTCs of patients exposed to radiation during childhood [10].

Several factors must be considered in the diagnostic, prognostic, and therapeutic landscape of differentiated thyroid carcinomas (DTCs) and medullary thyroid carcinoma (MTC). These include demographic (sex, age), clinical (symptomatology), laboratory (thyroglobulin levels), anatomopathological (tumor size, multifocality, extrathyroidal extension, lymphovascular invasion, presence of lymph node or distant metastases), and molecular factors [11,12].

Beyond previously discussed mutations, other molecular markers of potential prognostic interest include Pituitary Tumor Transforming Gene (PTTG), Ki-67%, and Galectin-3, which have been explored in preclinical studies, though real-world clinical correlation studies remain limited [13-17].

The protocol includes molecular and immunohistochemical analyses on tumor tissue samples, including archived paraffin-embedded specimens for a retrospective analysis and newly diagnosed cases with fresh paraffin samples. Additionally, the protocol incorporates previously collected molecular data, providing a comprehensive analysis of potential associations between molecular and histological features, clinical outcomes, and therapy response.

There remains a clear and unmet clinical need for novel prognostic and predictive biomarkers to better define thyroid cancer heterogeneity, improving classification and staging to guide prognosis and therapeutic decisions.

Thus, we have designed this study to collect and evaluate the clinical, laboratory, anatomopathological, and molecular characteristics of patients treated at the Medical Oncology Unit of the Fondazione Policlinico Universitario Agostino Gemelli (FPG) - IRCCS, both at diagnosis and during treatment, to investigate their prognostic and predictive value.

This objective aligns with FPG's recognition as an IRCCS for "Personalized Medicine" and as an Excellence Center recognized by the European Neuroendocrine Tumor Society (ENETS), making the study feasible given the high volume of patients with neuroendocrine neoplasms managed at the Medical Oncology Unit.

2. STUDY OBJECTIVES 2.1 Primary Objective

To evaluate the association between molecular markers (PTTG, Ki-67%, and Galectin-3) and survival outcomes, to assess their prognostic role in thyroid cancer patients across all disease stages.

2.2 Secondary Objectives

To correlate survival probability and treatment response with clinical, laboratory, anatomopathological, and molecular characteristics, identifying prognostic and predictive factors in thyroid cancer patients.

To evaluate duration of response (DoR), progression-free survival (PFS), disease control rate (DCR), and treatment tolerability (adverse events, AEs) across all therapy lines.

3. PATIENTS AND METHODS 3.1 Study Design

This is an observational, monocentric, ambispective study. It is spontaneous, not sponsored by pharmaceutical companies, and does not involve experimental drugs, devices, or procedures. The study includes immunohistochemical evaluation of Galectin-3 and molecular analysis of PTTG, which are not part of routine clinical practice. No additional costs will be incurred by the National Health System (SSN).

3.2 Study Population

The study includes patients with thyroid neoplasms followed at the Medical Oncology Unit of FPG - IRCCS. The study consists of:

Retrospective Cohort: Includes patients diagnosed or treated for thyroid cancer at FPG - IRCCS from January 1, 2010, until study approval.

Prospective Cohort: Includes patients newly diagnosed or starting thyroid cancer treatment at FPG - IRCCS for 60 months post-study approval.

4. STATISTICAL ANALYSIS

Descriptive analyses will be conducted on clinical, laboratory, radiological, anatomopathological, and molecular characteristics. Comparative analyses will be performed using Chi-square tests for categorical variables and Student's t-tests for continuous variables.

Cox proportional hazard models will estimate the relationship between variables and time-dependent endpoints (OS, PFS, and DoR). Kaplan-Meier survival curves will be plotted, and comparisons made using log-rank tests. Treatment tolerability will be assessed based on adverse event incidence (AEs).

Sample Size Calculation

Given the global incidence of thyroid cancer, an estimated sample size of ≥100 patients is considered feasible based on FPG - IRCCS enrollment capabilities.

5. ETHICAL CONSIDERATIONS

The study complies with:

Good Clinical Practice (GCP) guidelines Declaration of Helsinki Italian regulations on observational studies

Patient data will be anonymized and securely stored, following strict confidentiality protocols. The study will be approved by the Ethics Committee (EC) of FPG - IRCCS.

6. STUDY TIMELINE

Retrospective Cohort Data Collection: Approval - December 2023 Prospective Cohort Enrollment: Approval - February 2029 Data Analysis: March - May 2029 Publication & Presentation: June - September 2029

Estimated study duration: 60 months from Ethics Committee approval Projected completion date: September 2029

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of thyroid neoplasm, any subtype.
* Age ≥ 18 years.
* Signed informed consent (IC) for living patients.
* Signed data privacy consent for living patients.
* At least one follow-up visit after the initial oncology consultation.

Exclusion Criteria:

* Lack of clinical data sufficient to determine survival (primary endpoint of the study).
* Absence of a histological diagnosis.
* Failure to sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients diagnosed with thyroid neoplasms who are being followed at the Medical Oncology Unit of the Fondazione Policlinico Universitario Agostino Gemelli (FPG) - IRCCS. The study includes both a historical (retrospective) cohort and a prospective cohort.
  Retrospective Cohort: All patients diagnosed with thyroid cancer or who initiated treatment for thyroid cancer at the Medical Oncology Unit of FPG - IRCCS between January 1, 2010, and the date of study approval will be screened for enrollment.
  Prospective Cohort: All patients who receive a thyroid cancer diagnosis or initiate treatment at the Medical Oncology Unit of FPG - IRCCS during the 60 months following the study approval date will be screened for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2029-05-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | February 2025 - September 2029
  The time interval (expressed in months) between the date of disease diagnosis and the date of death from any cause.
  For patients who have not experienced an event by the date of the last follow-up, the observation period will be censored at that date.

SECONDARY OUTCOMES:
DoR, PFS, RR, DCR, Tolerability | February 2025 - September 2029
  DoR (Duration of Response): The interval between the first documented response and disease progression or death, whichever occurs first, expressed in months.
  PFS (Progression-Free Survival): The time elapsed from the start of treatment to disease progression or death, considering follow-up data, expressed in months.
  RR (Response Rate): The percentage of patients achieving a complete response (CR) or partial response (PR) according to RECIST 1.1 criteria.
  DCR (Disease Control Rate): The sum of CR, PR, and stable disease (SD) cases, expressed in percentage.
  Tolerability: Assessed by the incidence of adverse events (AEs), recorded according to CTCAE v5.0 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Schinzari, Prof, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS - UCSC, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sumana BS, Shashidhar S, Shivarudrappa AS. Galectin-3 Immunohistochemical Expression in Thyroid Neoplasms. J Clin Diagn Res. 2015 Nov;9(11):EC07-11. doi: 10.7860/JCDR/2015/16277.6760. Epub 2015 Nov 1. PMID 26673516